CLINICAL TRIAL: NCT05086016
Title: GROWTH: A Multicenter Pivotal Study of Neonatal, Infant, and Young Child Vascular Stenoses Studying the Renata Minima Stent
Brief Title: Growth Trial: Study of the Renata Minima Stent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renata Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC-0009
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Coarctation of the Aorta; Pulmonary Artery Stenosis
MeSH Terms: conditions — Aortic Coarctation; Stenosis, Pulmonary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All treated (Experimental): The All Treated (AT) population is defined as all subjects who signed informed consent, meet eligibility criteria and for whom a procedure was begun (defined as the initiation of vascular access with the Renata Minima system).
  Interventions: Device: Catheterized Stenting

INTERVENTIONS:
Device: Catheterized Stenting — Catheterized stenting of vascular narrowings.

SUMMARY:
The objective of the clinical investigation is to access clinical safety and effectiveness of the Minima Stent in neonates, infants, and young children requiring intervention for common congenital vascular stenosis (i.e., coarctation of the aorta and/or pulmonary artery stenosis) who are indicated for treatment.

ELIGIBILITY:
Inclusion criteria include:

* The subject's legally authorized representative has been informed of the nature of the clinical investigation, agrees to its provisions, and has provided written informed consent
* Requiring treatment* of:

  * native, acquired, or recurrent aortic coarctation, or
  * native, acquired, or recurrent pulmonary artery stenosis *As defined by the patient's medical team
* Patency of at least one femoral vein, femoral artery, jugular vein or both carotid arteries able to accommodate the delivery system
* Adjacent vessel to stenosis measuring > or equal to 4 mm

Exclusion criteria include:

* Active bloodstream infection requiring antibiotic therapy within 3 days prior to stent implantation
* History of or active endocarditis (active treatment with antibiotics) within 180 days prior to stent implantation
* Aortic or pulmonary artery aneurysm in the location targeted for treatment
* Body weight < 1.5 kg
* Anatomic location of lesion judged by the investigator to not lend to the safe placement of a stent
* Target vessels larger or smaller than the Minima System balloon size ranges
* Known genetic syndrome known to be associated with vasculopathies such as but not limited to Williams syndrome, Loeys-Dietz syndrome, etc
* Clinical scenario requiring that more than one vessel needs stent implantation at the time of the trial procedure.
* Currently participating in an investigational drug study or another device study
* Major or progressive non-cardiac disease resulting in a life expectancy of less than six months
* Known hypersensitivity to aspirin or heparin and cannot be treated with other antiplatelet and/or antithrombotic medications
* Known hypersensitivity to cobalt-chromium or contrast media that cannot be adequately pre-medicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2028-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Berman, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (7):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Boston Children's, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio
  - Le Bonheur Children's, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan PM, Zahn EM, Sathanandam S, Morray B, Shahanavaz S, Salavitabar A, Armstrong AK, Porras D, Berman DP. Multicenter Pivotal Trial of the Minima Stent for Vascular Stenosis in Infants and Young Children. Circ Cardiovasc Interv. 2025 Dec;18(12):e015618. doi: 10.1161/CIRCINTERVENTIONS.125.015618. Epub 2025 Oct 10. PMID 41070410

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Stent Implants
Period: Overall Study
Arm/Group | All Treated
Started | 42; 45 Stent Implants
Completed | 42; 45 Stent Implants (Of the 42 enrolled patients, 39 patients were treated with 1 Minima Stent and 3 patients with 2 Minima Stents, for a total of 45 Minima Stent Implants.)
Not Completed | 0; 0 Stent Implants

BASELINE CHARACTERISTICS:
Arm/Group | All Treated
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: months] | 9 [0.4 to 112]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 22
  More than one race | 0
  Unknown or Not Reported | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating Clinical Success at 6 Months
Description: The primary efficacy endpoint will be assessed as the rate of clinical success, with the performance goal defined as a clinical success rate of greater than 77%.
  Clinical success is defined as:
  * Stenosis relief, defined by stent outer diameter ≥ 75% of the surrounding vessel immediately after deployment.
  * Freedom from open surgical intervention required to treat Minima Stent disfunction through 6 months.
  * Maintenance of stented vessel diameter ≥ 50% of post-implant diameter at 6 months; as measured using CT angiography and/or angiography.
Time Frame: Through 6-month follow-up Visit
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 42
Participants | 41

2. Primary Outcome: Number of Participants With Freedom From Serious Adverse Events at 6 Months
Description: The primary safety endpoint will be assessed as the percentage of cases with freedom from procedure- or device-related SAEs resulting in an event listed below, with the performance goal defined as greater than 78% of cases:
  * Death
  * Cardiac arrest and/or emergency ECMO cannulation
  * Stroke
  * Limb loss
  * Vessel dissection of target lesion
  * Device thrombosis/occlusion
  * Cardiac perforation requiring percutaneous or open surgical intervention
  * Persistent cardiac arrhythmia requiring a pacemaker
Time Frame: Through 6-month follow-up Visit
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 42
Participants | 42

3. Secondary Outcome: Number of Patients With Arterial to Arterial Peak-to-peak Pressure Gradient of < 20 mmHg
Description: When a pressure gradient provides a reliable hemodynamic variable (e.g., coarctation of the aorta), a reduction in ventricle to arterial or arterial to arterial peak-to-peak pressure gradient to < 20 mmHg after stent placement.
Time Frame: immediately after deployment
Population: Patients with a Minima Stent deployed in the aortic circulation
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 21
Participants | 21

4. Secondary Outcome: Successful Stent Re-dilation at Re-catheterization
Description: Successful stent re-dilation (when indicated) at re-catheterization, defined as an increase in the intra stent angiographic luminal diameter within 2mm of the adjacent native vessel diameter immediately after re-dilation.
Time Frame: Immediately after re-dilation
Population: 15 patients have had at least one re-dilation with a total of 15 initial re-dilations and 6 second re-dilations (21 total re-dilations).
Measure: Count of Units; unit: Stent Re-Dilation Procedures
Units Other Than Participants: Stent Re-Dilation Procedures
Arm/Group | All Treated
Number analyzed (Participants) | 15
Number analyzed (Stent Re-Dilation Procedures) | 21
Stent Re-Dilation Procedures | 19

5. Secondary Outcome: Number of Patients With Freedom From Stent Embolization or Migration at 6 Months
Description: Freedom from stent embolization or migration through 6 months.
Time Frame: 6 months
Measure: Count of Units; unit: Stent Implants
Units Other Than Participants: Stent Implants
Arm/Group | All Treated
Number analyzed (Participants) | 42
Number analyzed (Stent Implants) | 45
Stent Implants | 42

6. Secondary Outcome: Number of Patients With Freedom From Stent Fracture at 6 Months
Description: Freedom from stent fracture that led to reintervention through 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 42
Participants | 42

7. Secondary Outcome: Number of Patients With Freedom From Non-elective Minima Stent Explant at 90-days Post Re-dilation
Description: Freedom from non-elective Minima Stent explant at 90-days post re-dilation procedure
Time Frame: 90 days post re-dilation
Population: 20 re-dilation procedures (14 post-initial re-dilation and 6 post-second re-dilation) across 14 subjects that have reached the 90 days post re-dilation procedure endpoint for assessment
Measure: Count of Units; unit: Stent Re-Dilation Procedures
Units Other Than Participants: Stent Re-Dilation Procedures
Arm/Group | All Treated
Number analyzed (Participants) | 14
Number analyzed (Stent Re-Dilation Procedures) | 20
Stent Re-Dilation Procedures | 20

8. Secondary Outcome: Number of Patients With Freedom From Procedure- or Device-related SAE During Re-dilation
Description: Freedom from procedure- or device-related SAE during re-dilation that results in the following:
  * Death
  * Cardiac arrest and/or emergency ECMO cannulation
  * Stroke
  * Limb loss
  * Vessel dissection of target lesion
  * Device thrombosis/occlusion
  * Cardiac perforation requiring percutaneous or open surgical intervention
  * Persistent cardiac arrhythmia requiring a pacemaker
Time Frame: Immediately after re-dilation
Measure: Count of Units; unit: Stent Re-Dilation Procedures
Units Other Than Participants: Stent Re-Dilation Procedures
Arm/Group | All Treated
Number analyzed (Participants) | 15
Number analyzed (Stent Re-Dilation Procedures) | 21
Stent Re-Dilation Procedures | 21

ADVERSE EVENTS:
Time Frame: Adverse Events are collected through study completion. Structured visits include at time of procedure, post-procedure/discharge, 1 month, 3 months, 6 months 12 months, and annually thereafter through 5 years.
Description: Serious Adverse Events are defined as procedure- or device-related SAEs resulting in an event of Death, Cardiac arrest and/or emergency ECMO cannulation, Stroke, Limb loss, Vessel dissection of target lesion, Device thrombosis/occlusion, Cardiac perforation requiring percutaneous or open surgical intervention, Persistent cardiac arrhythmia requiring a pacemaker.
  Adverse Events are defined as events related or possibly related to procedure or device
Arm/Group | All Treated
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 5/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated (N=42)
Access Site Complications (Injury, poisoning and procedural complications) | 5 (6) — Pulse Loss, Thrombus, Rebleed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT05086016/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT05086016/SAP_001.pdf